CLINICAL TRIAL: NCT03027765
Title: Prevalence of Constructed Space Maintainers in a Group of Egyptian Children Attending Pediatric Dentistry Department, Faculty of Oral and Dental Medicine Cairo University. A Cross-Sectional Study
Brief Title: Prevalence of Constructed Space Maintainers in a Group of Egyptian Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Abdelwahab AbdelHameed, Principle investigaror, Cairo University
Other Study IDs: Space Maintainers
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Egyptian children: Population1:
  Egyptian children with constructed space maintainers at Cairo University.
- Pediatric dentists: Population2:
  Pediatric dentists at Cairo University.

SUMMARY:
The purpose of the study is

* To determine the Prevalence of constructed space maintainers at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.
* To assess the knowledge, attitude and awareness of constructed space maintainers for pediatric patients' guardians at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

and

- To assess the knowledge, attitude and practice of pediatric dentists towards use of space maintainers in children, at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

DETAILED DESCRIPTION:
The purpose of the study is

* To determine the Prevalence of constructed space maintainers at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.
* To assess the knowledge, attitude and awareness of constructed space maintainers for pediatric patients' guardians at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

and

- To assess the knowledge, attitude and practice of pediatric dentists towards use of space maintainers in children, at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

PO1:

Population:

Egyptian children with constructed space maintainers and their guardians attending Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

Outcome1:

Prevalence of constructed space maintainers Knowledge, attitude and awareness of constructed space maintainers for pediatric patients' guardians.

PO2

Population2:

Pediatric dentists at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.

Outcome2:

knowledge, attitude and practice of pediatric dentists towards the use of the space maintainers.

ELIGIBILITY:
i have two population

1st population is Pediatric patients

Inclusion criteria for pediatric patients:

1. All patients with constructed space maintainers
2. Positive patient's acceptance for participation in the study.
3. Both genders are included.
4. Children Medically free from any systemic disease.

Exclusion criteria for pediatric patients:

1. Patients with orthodontic appliances.
2. Patient having one of the different following habit thumb sucking, lip biting, tongue thrusting etc.

2nd population is pediatric dentists:

Inclusion criteria for Pediatric dentists:

-All Pediatric dentists having master degree and above.

Exclusion criteria for Pediatric dentists:

-Pediatric dentists refused to participate in the study.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian children with constructed space maintainers and their guardians attending Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University Both gender are included and Pediatric dentists at Pediatric Dentistry and Dental Public Health Department, Faculty of Oral and Dental Medicine, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of constructed space maintainers | 6 months
  Device for measurement through Visual examination and unit is Binary (Yes, No) and MCQ

CONTACTS AND LOCATIONS:
Overall Officials: Sherine Ezz Eldin Taha, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ari T. Follow-up problems with fixed appliances in pediatric dentistry. N Y State Dent J. 2015 Mar;81(2):16-20. PMID 25928968
- [Background] Asiry MA. Occlusal Status among 12-16 Year-Old School Children in Riyadh, Saudi Arabia. J Int Oral Health. 2015 May;7(5):20-3. PMID 26028897
- [Background] Baroni C, Franchini A, Rimondini L. Survival of different types of space maintainers. Pediatr Dent. 1994 Sep-Oct;16(5):360-1. No abstract available. PMID 7831141
- [Background] Brothwell DJ. Guidelines on the use of space maintainers following premature loss of primary teeth. J Can Dent Assoc. 1997 Nov;63(10):753, 757-60, 764-6. PMID 9401297
- [Background] Dhar V, Jain A, Van Dyke TE, Kohli A. Prevalence of gingival diseases, malocclusion and fluorosis in school-going children of rural areas in Udaipur district. J Indian Soc Pedod Prev Dent. 2007 Apr-Jun;25(2):103-5. doi: 10.4103/0970-4388.33458. PMID 17660647
- [Background] Dogan MC, Dogan SK, Kendi E. Complications of pediatric denture misuse: a case report. Oral Health Prev Dent. 2005;3(2):127-30. PMID 16173390
- [Background] Green J. Mind the gap: Overview of space maintaining appliances. Dent Nurs 2015; 11(1):24-7.
- [Background] Kapala JT. Interceptive orthodontics and management of space problems. In: Braham RL, Morris ME. Textbook of Pediatric Dentistry, Eds. Baltimore, London, William & Wilkins Co. 1980: pp 320-356.
- [Background] Keski-Nisula K, Hernesniemi R, Heiskanen M, Keski-Nisula L, Varrela J. Orthodontic intervention in the early mixed dentition: a prospective, controlled study on the effects of the eruption guidance appliance. Am J Orthod Dentofacial Orthop. 2008 Feb;133(2):254-60; quiz 328.e2. doi: 10.1016/j.ajodo.2006.05.039. PMID 18249292
- [Background] Laing E, Ashley P, Naini FB, Gill DS. Space maintenance. Int J Paediatr Dent. 2009 May;19(3):155-62. doi: 10.1111/j.1365-263X.2008.00951.x. PMID 19385999
- [Background] Leite-Cavalcanti A,de Alencar, Benzerra PK,Garcia A., Prevalence of early loss of primary molars in school children in Brazil. Pak Oral Dent J 2008; 28:113-6.
- [Background] Petrunov V. Epidemiological research of malocclusions and the need of orthodontic treatment among the Bulgarians in the mixed to permanent dentition period, Disertation, Sofia 2012, p.62
- [Background] Qudeimat MA, Fayle SA. The use of space maintainers at a UK pediatric dentistry department. ASDC J Dent Child. 1999 Nov-Dec;66(6):383-6. PMID 10656119
- [Background] Ronnerman A, Thilander B. A longitudinal study on the effect of unilateral extraction of primary molars. Scand J Dent Res. 1977 Jul;85(5):362-72. doi: 10.1111/j.1600-0722.1977.tb01516.x. PMID 268677
- [Background] Ronnerman A, Thilander B. Facial and dental arch morphology in children with and without early loss of deciduous molars. Am J Orthod. 1978 Jan;73(1):47-58. doi: 10.1016/0002-9416(78)90101-x. No abstract available. PMID 271472
- [Background] Talekar BS, Rozier RG, Slade GD, Ennett ST. Parental perceptions of their preschool-aged children's oral health. J Am Dent Assoc. 2005 Mar;136(3):364-72; quiz 381. doi: 10.14219/jada.archive.2005.0179. PMID 15819352